CLINICAL TRIAL: NCT04924244
Title: Effect of Music on Pain and Anxiety in Chronic Pain Patients Undergoing Lumbar Interventional Procedures
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Milton S. Hershey Medical Center (Other)
Responsible Party: Principal Investigator, Bunty Shah, Assistant Professor of Anesthesiology & Perioperative Medicine, Milton S. Hershey Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 16112
Record Dates: First submitted 2021-06-07; First posted 2021-06-11 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2025-10

CONDITIONS: Chronic Pain; Anxiety
MeSH Terms: conditions — Chronic Pain; Anxiety Disorders | interventions — Music Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- No Music (Active Comparator): No music will be played during the subject's standard of care lumbar spinal interventional procedure (including: epidural steroid injections, facet injections, medial branch blocks).
  Interventions: Other: No Music
- Music Therapy (Experimental): Music of the subject's preferred genre will be played during the subject's standard of care lumbar spinal interventional procedure (including: epidural steroid injections, facet injections, medial branch blocks).
  Interventions: Other: Music Therapy

INTERVENTIONS:
Other: Music Therapy — We will play music of the subject's choice of genre during the procedure.
  Arms: Music Therapy
Other: No Music — No music will be played during the subject's interventional procedure
  Arms: No Music

SUMMARY:
The purpose of this study is to evaluate, subjectively and objectively, whether playing music during procedures for treatment of chronic lower back pain has an effect on patients' anxiety and pain. The investigators hypothesize that playing music will result in reduced patient reported anxiety and pain scores and less variation from baseline of vital signs versus patients in the control group without music therapy. This is a pilot study.

ELIGIBILITY:
Inclusion Criteria:

1. Age greater than or equal to 18
2. Female or male
3. Patients undergoing standard of care lumbar spinal interventional procedures including: epidural steroid injections, facet injections, medial branch blocks

Exclusion Criteria:

1. Patients who cannot consent for themselves, including cognitively impaired patients.
2. Non-English speaking patients
3. Patients taking beta blocker medication
4. Patients that have a pacer and have a set rate
5. Patients with self-reported hearing problems or with hearing aids

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2021-07-15 (Actual); Primary Completion 2026-02-28 (Estimated); Study Completion 2026-02-28 (Estimated)

PRIMARY OUTCOMES:
Pre-procedure State-Trait Anxiety Inventory (STAI) Score | Within 30 minutes prior to the subject's interventional procedure
  A measure of anxiety in a person. Higher score correlates increased anxiety and worsened outcome. The minimum score is 40 and the maximum score is 160.
Post-procedure State-Trait Anxiety Inventory (STAI) Score | Within 30 minutes following to the subject's interventional procedure
  A measure of anxiety in a person. Higher score correlates with increased anxiety and worsened outcome. The minimum score is 40 and the maximum score is 160.

SECONDARY OUTCOMES:
Pre-procedural Visual Analog Score (VAS) for pain | Within 30 minutes prior to the subject's interventional procedure
  Visual Analog Score for pain. Higher score correlates with increased pain and worsened outcome. The minimum score is 0 and the maximum score is 10.
Post procedural Visual Analog Score (VAS) | Within 30 minutes following the subject's interventional procedure
  Visual Analog Score for pain. Higher score correlates with increased pain and worsened outcome. The minimum score is 0 and the maximum score is 10.

CONTACTS AND LOCATIONS:
Overall Officials: Bunty Shah, Principal Investigator — Milton S. Hershey Medical Center
Locations (1):
- Milton S. Hershey Medical Center, Hershey, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No